CLINICAL TRIAL: NCT03646006
Title: A Randomized Controlled Trial (RCT) Comparing Presacral Nerve Block Versus Sham Block on Post-operative Pain in Women Undergoing Total Laparoscopic Hysterectomy.
Brief Title: The Effect of Pre-sacral Nerve Block on Immediate Post-operative Pain Following Laparoscopic Hysterectomy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Mara Sobel, Assistant Professor, Core Obstetrics and Gynecology, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSH REB 16-0203-A
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-sacral nerve block (Experimental): 10 mL bupivacaine (5mg/mL)
  Interventions: Drug: Bupivacaine
- Sham block (Sham Comparator): 10 mL normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — 10 mL (5mg/mL)
  Arms: Pre-sacral nerve block
Drug: Placebo — 10 mL normal saline
  Arms: Sham block

SUMMARY:
Hysterectomy (removal of the uterus) is the most common major gynecologic surgery performed in Canada. With a focus on minimally invasive techniques and optimization of peri-operative pain control, gynaecologists have made great strides towards reducing hospital stay and accelerating post-operative recovery. These are essential achievements, both for patients and their families and for our resource-limited public healthcare system.

Optimization of peri-operative pain control is multifactorial and includes, for example, administration of pre-operative analgesics, infiltration of incision sites with local anesthetic and provision of post-operative pain medications. As the understanding of pain mechanisms evolves, the incorporation of intra-operative nerve blocks has become yet another effective strategy to reduce post-operative pain.

The presacral nerve plexus, which carries nerve fibers from the uterus to the brain, is an important pathway that transmits midline pelvic pain in women. Destruction of the pre-sacral nerves has been shown to provide excellent pain control in a variety of clinical settings.

While transection of the presacral nerve at the time of surgery is technically challenging, instilling a presacral nerve block is surprisingly straightforward making this technique safe to perform in the hands of many gynecologists. In this technique, local anesthetic is instilled into the presacral space using a needle inserted through the abdomen.

Given that the presacral nerve plexus is an integral pain pathway for the uterus, the investigators hypothesize that the addition of a presacral nerve block during laparoscopic (camera surgery) hysterectomy would confer an additional reduction in immediate post-operative pain. The proposed study therefore aims to look at the impact of presacral nerve block versus a sham (blank) block on immediate post-operative pain in a group of women scheduled to undergo laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to determine the effectiveness of a presacral nerve block on post-operative pain following total laparoscopic hysterectomy. Given that the presacral nerves carry pain sensation from the midline pelvic structures suggests that blocking this important nerve pathway intra-operatively would provide an excellent complementary method of analgesia in this patient population. Considering the frequency of hysterectomy, further improvements in pain management with this simple additional step could offer great benefits for patients and for the healthcare system by minimizing narcotic consumption, hospital stay, recovery time and time away from work.

Methodology:

This study is a single-center parallel group randomized controlled trial (RCT) comparing the administration of a presacral nerve block using 10 millilitres (mL) of local bupivacaine (5 milligrams [mg]/ml) versus 10 mL of normal saline (sham block). Participants will be selected using a convenience sample from Mount Sinai Hospital's outpatient gynecology clinics. All women undergoing total laparoscopic hysterectomy will be considered for this study. Baseline characteristics, including age, gravity, parity, medical history, surgical history, body mass index (BMI) and indication for surgery will be collected on all study participants.

Study participants will be randomized on the day of surgery. The investigators will create a randomization list using a computer-generated allocation sequence in equal ratio. The investigators will place the drug/placebo designation in numbered opaque envelopes and secure the envelope to the patient's chart on the day of surgery. The randomization number will correspond to a pre-filled syringe (containing either drug or placebo) that will be labelled with the randomization number only. A list of syringe numbers and corresponding group allocation will be kept on a secured server and will not be visible to the surgeon or study personnel. The surgeon will complete the laparoscopic hysterectomy according to his/her preferred operative technique. After the hysterectomy is completed, and prior to desufflating the abdomen, the surgeon will be presented with study drug (bupivicaine/placebo) loaded in a syringe with a spinal needle. The surgeon will laparoscopically instill the drug/placebo into the presacral space after confirming hemostasis as the final step before closing the abdomen.

The surgeon, research team, participants and data analysts will be blinded to treatment group. Participants will receive standard perioperative care including induction/maintenance of general anesthesia and prevention/treatment of post-operative nausea, vomiting and pain. Following surgery, patients will complete a self-administered visual analogue scale [VAS] for pain at 1-, 2- and 3-hours after surgery (primary outcome). In addition, the investigators will calculate total narcotic and anti-emetic consumption prior to discharge and report on any adverse events (secondary outcomes).

Outcomes:

The primary outcome will be early post-operative pain measured at 3-hours following surgery by a self-administered VAS for pain. Secondary outcome measures will include: (a) pain measured at 1- and 2-hours following surgery by a self-administered VAS for pain (b) total narcotics administered from end of surgery until discharge and (c) adverse effects/complication rates. The following will also be collected: estimated blood loss; operative time; total length of stay in post-anaesthesia recovery unit (PACU) prior to discharge; time to first void after surgery; and time to first ambulation after surgery. Due to the short follow up period for the majority of data collection, the investigators anticipate near 100% retention of study subjects.

Statistics:

Based on a sample-size calculation to detect a 30% reduction in self-reported pain using a VAS for pain (with alpha 0.05 and power 0.9) the study will require 30 patients per group. With a conservative estimate of 5 total laparoscopic hysterectomies per week, the investigators expect to surpass this target within 6 months of starting our study.

Success of the intervention will be assessed by comparing primary and secondary outcome measures between the two treatment arms using an independent student T-test (α = 0.05) for continuous variables and expressed as the difference between means with accompanying 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective total laparoscopic hysterectomy
* Age > 18 years

Exclusion Criteria:

* Previous presacral neurectomy
* Concurrent surgical procedure other than salpingectomy and/or oophorectomy
* Gynecological cancer beyond stage 1 disease
* Chronic narcotic consumption
* Fibromyalgia
* Inability to provide consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain at 3 hours | 3 hours post-operatively
  Pain measured on a visual analogue scale (VAS). Range will be from zero (no pain) to 10 (most pain).

SECONDARY OUTCOMES:
Post-operative pain at 1 hour | 1 hour post-operatively
  Pain measured on a visual analogue scale (VAS). Range will be from zero (no pain) to 10 (most pain).
Post-operative pain at 2 hours | 2 hours post-operatively
  Pain measured on a visual analogue scale (VAS). Range will be from zero (no pain) to 10 (most pain).
Post-operative narcotic consumption | On day of surgery
  Total dose of narcotics consumed by the patient from end of surgery (time of extubation) until time of discharge
Post-operative anti-emetic consumption | On day of surgery
  Total dose of anti-emetics consumed by the patient from end of surgery (time of extubation) until time of discharge
Adverse Events | 6 weeks following surgery
  Any adverse events described during the operation, in the post-anaesthesia care unit (PACU) or reported by the patient at the 6-week post-operative visit.

OTHER OUTCOMES:
Estimated blood loss | On day of surgery
  Amount of blood lost during the surgery (as reported by the surgical team)
Operative Time | On day of surgery
  Duration of surgery (from first skin incision to time of extubation)
Time to first ambulation | On day of surgery
  Duration of time from end of surgery (time of extubation) until first ambulation
Time to first void | On day of surgery
  Duration of time from end of surgery (time of extubation) until first urination
Time to discharge | On day of surgery
  Total duration of time between end of surgery (time of extubation) until discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Mara Sobel, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No